CLINICAL TRIAL: NCT06124742
Title: Alteration of Taste Among Orthodontic Patients Following Clear Aligners Treatment: A Prospective Cohort Study
Brief Title: Alteration of Taste Among Orthodontic Patients Following Clear Aligners Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Sponsor
Other Study IDs: FPGRP/2023/722/949/888; Riyadh Elm University (Other: February 2004)
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-06

CONDITIONS: Taste Perception; Orthodontic Appliance Complication; Fixed Orthodontic Appliances
Keywords: Orthodontic Appliance; Taste Perception; clear aligners

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- clear aligners: The aim of this study is to assess the gustatory perception and alteration in patients using either clear aligners or fix orthodontics treatment.
  Interventions: Device: clear aligners

INTERVENTIONS:
Device: clear aligners — taste perception will be evaluated before and after using clear aligners.

SUMMARY:
The goal of this clinical trial is aimed to assess the gustatory perception and alteration in patients using either clear aligners or fix orthodontics treatment in orthodontic patient aged +18 years and not have any endocrine abnormalities, internal diseases, middle ear affections, xerostomia, or depression.

The main question it aims to answer are:

Does the clear aligner have an effect on taste perception following the treatment? Participants will be given a questionnaire before and after the orthodontic treatment to assess the taste perception following the orthodontic treatment. In addition, The Burghart taste strips (ODOFIN taste strips) will clinically assess the taste's function by using four concentrations on three separate occasions (T0, T1, and T2) ,The taste strips will be placed in about the same order; they will apply to the protruding tongue immediately posterior to its first third, either to the left or right side, to study lateralization. subjects will then be asked to close their mouths and choose one of five possible answers on a scale (sweet, sour, salty, bitter, no taste).

DETAILED DESCRIPTION:
In Saudi Arabia, one of the common oral health problems is the malocclusion. Crowding was the commonest type of malocclusion followed by increased spacing and overjet (Al-Hummayan, 2018). Malocclusion prevalence varies among different populations globally based on multiple factors including the time of the study, the geographical location. In addition , the selection criteria used for the sample selection, such as age and gender, are all factors that contribute to the malocclusion . Profitt, 2005 reported that 57-59% of Americans had at least some orthodontic treatment needed (Profitt WR, 1998). In the UK, the percentage was 59% (Foster TD, 1974), and in Jordan, it was 92% (Abu Alhaija ES, 2005 ) . There was a report that 40%-62% of Saudi Arabia needed orthodontic treatment (Baseer MA, 2021).

Clear aligner is an alternative to traditional braces that helps to guide the teeth into their proper positions. Unlike braces, clear aligners control tooth movement without metal weirs or brackets. All aligners made of strong plastic materials and made to fit each individual's mouth. the alignment of the teeth can be accomplished using a series of aligners in which each aligner moves the teeth incrementally until the desired result is achieved (Tigani, n.d.).

Orthodontics treatment aims to improve patient quality of life by improving both function and appearance of teeth. So, treatment complications during the treatment plan must be addressed. One of the most important things is proper taste perception. impaired perception of taste stimuli may occur as a result of a foreign body such as placement of the orthodontic material in the oral cavity (Izabella Dunin-Wilczyńska1, 2011).

Through the literature review, many studies were performed on alteration in taste sensation with using removable appliances, and all results were statistically not significant (Hegde AM, 2007) (Sarawan Siripanthana D.D.S., 2015) (Razdan P, 2017). A study analysed the change in taste perception in children using removable orthodontic appliances by using different taste stimuli and asking the children to score as per their perception. There was no statistically significant difference between the study and control groups (Razdan P, 2017). Moreover, a further investigation was conducted on patients who received upper removable orthodontic devices with posterior bite planes, and they used the Modified Harris-Kalmus test to measure the four tastes. salty, sweet, bitter, and sour. this study showed no effect on the taste recognition threshold of the four taste qualities, according to the results of this study (Sarawan Siripanthana D.D.S., 2015). However, alterations of taste perception in orthodontic patients are not studied sufficiently.

Taste is considered a multisensory experience (Shaikh & Soni., 2022), which contains five senses of taste salty, sour, bitter, sweet, and umami, the last being the Japanese term for a savoury sensation (J., 2004). Gustation loss may arise due to a diverse spectrum of systemic or acute clinical conditions or medications. Moreover, a published article done by otolaryngologists used taste strips, and the results of the study indicate the usefulness of the taste strips in a clinical context (Mueller C, 2003). So based on this article will use the strips which are made from filter paper and impregnated with different taste solutions. taste disturbance can also reduce the pleasure of life and cause a significant reduction in patients' quality of life. It is important, therefore, the main aim of this study to evaluate taste perception following the orthodontics treatment.

To the best of author's knowledge, no study has been published to assess taste perception and taste change after clear aligners treatment. Using clear aligners treatment, the present study aims to assess the effect of taste perception and alteration on taste perception and perception.

Literature review:

Taste perception in orthodontics patients has insufficient studies. There are two studies done on taste perception in patients wearing a removable orthodontic appliance. There are various complaints known related to a removable orthodontic appliance. A study done over 100 volunteers aged between (8-13 years old) to evaluate the complaint regarding appliances and their effect on taste and flavor perception, was divided into two groups (I and II) of 50 children each being divided as study and control groups. Selected volunteers were given samples consisting of eight different taste and flavor stimuli and were asked to score as per their perception in different testing sessions. The overall results revealed that volunteers from both study and control groups, irrespective of the use of removable orthodontic appliances showed marked variation in the estimation of the taste and flavor stimuli in different testing sessions. However, the results obtained were statistically not significant (Hegde AM, 2007).

One short-term study was comparing the recognition of the four taste qualities in Eighteen young patients aged (8-14 years old) wearing upper removable orthodontic appliances with posterior bite planes before and after insertion by using Modified Harris-Kalmus test. The analyses were conducted using SPSS, both Friedman test and Test-retest reliability were used, and the results showed no significant differences (Sarawan Siripanthana D.D.S., 2015).

Another study aimed to analyze the taste perception in 100 young children aged (8- 13 years old) undergoing upper removable orthodontic appliance therapy. the study was divided into two groups (groups I and II) of 50 children each as study and control groups. They used eight different taste stimuli samples consisting of 5 mL samples representing tasteless, sweet, salty, and sour substances. Using verbal score and visual analog scale, the scoring of the volunteers was nearly constant, indicating that an appliance does not play a major role in the alteration of taste stimuli (Razdan P, 2017).

Aim of the research:

The aim of this study is to assess the gustatory perception and alteration in patients using either clear aligners or fix orthodontics treatment.

Specific Objectives:

* To analyze the complaint regarding clear appliances and their effect on taste and flavor perception.
* To quantitatively evaluate taste perception by using taste strip.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in orthodontic therapy using either clear aligners or fixed orthodontic treatment.
2. Healthy patients aged 18 years and over.

Exclusion Criteria:

1. endocrine abnormalities (thyroid gland dysfunction, diabetes mellitus, Cushing's disease).
2. internal diseases (chronic renal failure, liver cirrhosis).
3. middle ear affections.
4. xerostomia.
5. depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is a prospective cohort study. The study will be carried out at Riyadh Elm university clinic. The investigation will involve 134 participants (aged variety from 15 to 40 years old). A self-administrated questionnaire will be used before and after the orthodontic treatment to assess the taste perception following the clear aligners treatment. In addition, The Burghart taste strips (ODOFIN taste strips) will use clinically to evaluate the taste perceptions.
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
assess the gustatory perception and alteration in patients using either clear aligners or fix orthodontics treatment. | On three separate occasions, the testing procedures will be carried out. - T0- one month before the appliance is installed. - T1- immediately after appliance installation. - T2- six months after appliance installation.
  - To analyze the complaint regarding clear appliances and their effect on taste and flavor perception. - To quantitatively evaluate taste perception by using taste strip.

CONTACTS AND LOCATIONS:
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alhummayani FM, Taibah SM. Orthodontic treatment needs in Saudi young adults and manpower requirements. Saudi Med J. 2018 Aug;39(8):822-828. doi: 10.15537/smj.2018.8.22337. PMID 30106421
- [Background] Proffit WR, Fields HW Jr, Moray LJ. Prevalence of malocclusion and orthodontic treatment need in the United States: estimates from the NHANES III survey. Int J Adult Orthodon Orthognath Surg. 1998;13(2):97-106. PMID 9743642
- [Background] Foster TD, Day AJ. A survey of malocclusion and the need for orthodontic treatment in a Shropshire school population. Br J Orthod. 1974 Apr;1(3):73-8. doi: 10.1179/bjo.1.3.73. No abstract available. PMID 4525734
- [Background] Abu Alhaija ES, Al-Khateeb SN, Al-Nimri KS. Prevalence of malocclusion in 13-15 year-old North Jordanian school children. Community Dent Health. 2005 Dec;22(4):266-71. PMID 16379166
- [Background] Baseer MA, Almayah NA, Alqahtani KM, Alshaye MI, Aldhahri MM. Oral Impacts Experienced by Orthodontic Patients Undergoing Fixed or Removable Appliances Therapy in Saudi Arabia: A Cross-Sectional Study. Patient Prefer Adherence. 2021 Dec 2;15:2683-2691. doi: 10.2147/PPA.S343084. eCollection 2021. PMID 34880603
- [Background] Hegde AM, Dwivedi S. Effect of removable orthodontic appliance on taste and flavor perception--a clinical study. J Clin Pediatr Dent. 2007 Fall;32(1):79-82. doi: 10.17796/jcpd.32.1.jt1677554845122u. PMID 18274477
- [Background] Razdan P, Sakthivel VS, Naqvi ZA, Goyal V, Tripathi S, Singh S. Alteration in Taste Perception among Young Children during the use of Removable Orthodontic Appliance Therapy. J Contemp Dent Pract. 2017 Jul 1;18(7):607-613. doi: 10.5005/jp-journals-10024-2093. PMID 28713117
- [Background] Bradbury J. Taste perception: cracking the code. PLoS Biol. 2004 Mar;2(3):E64. doi: 10.1371/journal.pbio.0020064. Epub 2004 Mar 16. PMID 15024416
- [Background] Mueller C, Kallert S, Renner B, Stiassny K, Temmel AF, Hummel T, Kobal G. Quantitative assessment of gustatory function in a clinical context using impregnated "taste strips". Rhinology. 2003 Mar;41(1):2-6. PMID 12677732